CLINICAL TRIAL: NCT05574309
Title: Understanding the Measurement of Girdle Dissociation in the Fall of the Older People Subject. Case-control Study
Brief Title: Understanding the Measurement of Girdle Dissociation in the Fall of the Older People Subject.
Acronym: EPAD-C2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21CH030; ANSM (Other: 2022-A00796-37)
Record Dates: First submitted 2022-10-03; First posted 2022-10-10 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-04

CONDITIONS: Fall Patients; Frailty
Keywords: fall prevention; older; inertial sensors; dissociation of girdles
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: Case-control study from the clinical gerontology service and the PROOF cohort. Cases: patients who fell (= at least one fall in the last 12 months) mainly from the clinical from the clinical gerontology department.
  Controls: patients/subjects who have not fallen, mainly from the PROOF cohort.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fallers (Sham Comparator): population of patients who have fallen from the clinical gerontology department of the CHU of Saint-Etienne and from the PROOF cohort and subjects of the Office Stéphanois pour les Ainés (OSAP)
  Interventions: Device: Dissociation measure of pelvic and scapular girdles by inertial sensors of accelerometer; Device: GAITRite Device
- non fallers (Other): population of patients who did not fall from the clinical gerontology department of the CHU of Saint-Etienne and from the PROOF cohort and subjects of the Office Stéphanois pour les Ainés (OSAP)
  Interventions: Device: Dissociation measure of pelvic and scapular girdles by inertial sensors of accelerometer; Device: GAITRite Device

INTERVENTIONS:
Device: Dissociation measure of pelvic and scapular girdles by inertial sensors of accelerometer — Dissociation measure of pelvic and scapular girdles by 2 inertial sensors of accelerometer type (IMU BNO055) during a 10 m walking test
Device: GAITRite Device — Walking parameter measured during a 10 m walking test with GaitRite device

SUMMARY:
Falls, especially in the older people, are frequent with potential serious consequences. The strategy for preventing falls involves detecting the fall risk. Current tests to determine the risk of falling are too late indicators of gait disorder. Loss of gait dissociation is an element associated with the mechanism of the fall and appears earlier. Its diagnosis is particularly important as it is a reversible impairment if rehabilitation interventions can be proposed to correct this anomaly.

DETAILED DESCRIPTION:
The purpose of this study is to validate the device's measurement of belt dissociation in a discriminating manner between fallers and nonfallers.

ELIGIBILITY:
Inclusion Criteria:

* Informed and signed a written consent form.
* Affiliated or eligible to a health insurance system.
* Being able to give their consent to participate.
* For fallers: had at least one fall in the previous year.
* For non fallers: not had a fall in the previous year.

Exclusion Criteria:

* Patients suffering from a neurological or articular pathology responsible for gait disorders (Parkinson's disease, hemiplegia, narrow lumbar canal, peripheral neuropathy, vestibular pathology, chronic inflammatory rheumatism…).
* Patients who have undergone joint surgery of the lower limbs during the year.
* Patients walking with a walker.
* Patients with an internal electronic device (pacemaker, neurostimulator, insulin pump…).
* Patients taking long-term neuroleptics.
* Patients with advanced major cognitive impairment (according to the Clinical Dementia Rating Protocol >1).

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 112 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2025-01-17 (Actual)

PRIMARY OUTCOMES:
measure of position of the pelvic and scapular girdles | During walking test
  The position of the pelvic and scapular girdles will be measured by the angle (in degrees) between the two girdles C7 and L5 in the sagittal plane during a 10 meters walking test. The angle will be measured by two inertial sensors of accelerometer type (IMU BNO055).

SECONDARY OUTCOMES:
assessment of patients' frailty status | at the inclusion
  Patients' frailty status will be assessed using the Fried score
assessment of patients' frailty status | During walking test
  Patients' frailty status will be assessed using the Fried score
Composite outcome : measurement of various walking quantitative parameters | at the inclusion
  Composite outcome will be measured with the following quantitative parameters using the GAITRite device: the parameters of walking speed (m/s), variability (%), length (m), width (cm), symmetry (m), cadence (steps/min) and step cycle time (s).
Composite outcome : measurement of various walking quantitative parameters | During walking test
  Composite outcome will be measured with the following quantitative parameters using the GAITRite device: the parameters of walking speed (m/s), variability (%), length (m), width (cm), symmetry (m), cadence (steps/min) and step cycle time (s).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas CELARIER, PhD, Principal Investigator — Centre Hospitalier Universitaire de Saint Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No